CLINICAL TRIAL: NCT07275203
Title: Concordance of the Biology of Primary Breast Carcinoma and the Biology of Recurrence , Retrospective Study.
Brief Title: Concordance of the Biology of Primary Breast Carcinoma and the Biology of Recurrence .
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mera Samy George Samy, Principle Investigator, Sohag University
Other Study IDs: Soh-Med--25-11-8MS
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-11

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
the study will discuss the concordance of the biology of primary breast carcinoma and the biology of recurrence.

The study will be conducted at Department of Clinical Oncology, Sohag University Hospital and Sohag Cancer center, Sohag, Egypt.

including Patients diagnosed and treated between 2015 and 2025 and Data will be collected from medical records, pathology reports, and radiology reports.

ELIGIBILITY:
Inclusion Criteria:

* Age more than18 years old at time of diagnosis of breast cancer.
* Patients who had recurrent breast cancer following adjuvant treatment.
* Biopsy was taken from the site of recurrence and biology was done.

Exclusion Criteria:

* Patients with distant metastasis at time of presentation.
* Patients diagnosed with double malignancy.
* Patients with incomplete data records.
* Recurrent breast cancer and biopsy difficult to be taken .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted at Department of Clinical Oncology, Sohag University Hospital and Sohag Cancer center, Sohag, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Rate of receptor discordance between primary and recurrent breast cancer. | 2015-2025